CLINICAL TRIAL: NCT06208163
Title: Psychoneuroimmunology as a Framework for Studying the Effects of Chiropractic Care in a Population With High Central Adiposity: a Feasibility Trial
Brief Title: The Effects of Chiropractic in a Population With High Central Adiposity
Acronym: OBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Life University (Other)
Collaborators: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-0027
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-02

CONDITIONS: Abdominal Obesity
Keywords: abdominal obesity; adults; psychoneuroimmunology; chiropractic
MeSH Terms: conditions — Obesity, Abdominal | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chiropractic care (Experimental): 6 weeks of chiropractic care
  Interventions: Procedure: Chiropractic

INTERVENTIONS:
Procedure: Chiropractic — Chiropractic spinal adjustments

SUMMARY:
Since 1980, the global prevalence of obesity, commonly defined as a body mass index (BMI) of 30 or higher, has doubled. Importantly, high levels of central adiposity (i.e., abdominal fat) is associated with numerous PNI-related sequelae, including increased levels of psychological distress, cognitive deficits, ANS dysfunction, and immune marker abnormalities. To our knowledge, rigorous investigation of chiropractic's impact on psychoneuroimmunological (PNI)-related outcomes in people with high central adiposity is lacking. Based on limited evidence to date, it is plausible that clinically important PNI-related dysfunctions (e.g., heightened stress levels, executive function impairments, dysautonomia, immune dysregulation) common in this population could be ameliorated via chiropractic care.

DETAILED DESCRIPTION:
Up to twenty (20) obese individuals (18-65 yrs of age) will be recruited. For our trial, obesity will be indexed as a BMI ≥30 and an elevated waist circumference (i.e., >35 inches for women, >40 inches for men).

Subjects will be asked to do the following…

* Restrict certain behaviors prior to their lab visits which include 1) 3 hours prior abstain from caffeine, brushing your teeth, alcohol-based mouthwash, nicotine, food, & drinking large amounts of liquid very quickly (e.g., chugging a 16 oz bottle of water; sipping water is ok) and 2) 24 hours prior abstain from strenuous exercise, alcohol, & over the counter drugs (e.g., antihistamines, Tylenol, etc.)
* Have their height, weight, and waist circumference measured.
* Drool into a tube for subsequent testing of immune markers (i.e., salivary IgA)
* Have electrodes placed on/around their chest & back to measure respiration, ECG, and impedance cardiography (ICG)
* Perform a postural challenge whereby they lay supine (8 min), stand quickly (3 min), and return quickly to the supine position (3 min).
* Have their cognitive function assessed while walking on a treadmill (dual task).
* Answer questions about their mental, physical, and emotional health.
* Receive 6-weeks of chiropractic adjustments from community-based clinicians.

Assessments will take place at baseline, after 2 weeks of chiropractic, and after 6 weeks of chiropractic.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Body mass index (BMI) at least 30
* Waist circumference at least 35 inches if female or 40 inches if male

Exclusion Criteria:

* Had chiropractic care within the past 30 days
* Prescribed short-acting benzodiazepines which include midazolam & triazolam
* If taking prescription medications, other than short-acting benzodiazepines, not on a stable dose for a minimum of 6 weeks with plans to change medications or doses during the study
* Not able to walk unassisted on a treadmill
* Known disorder resulting in syncope/fainting during postural changes (e.g., POTS, orthostatic hypotension)
* Pacemaker or known heart condition that influences the electrical or mechanical function of the heart (e.g., severe heart valve disease)
* Diagnosed with externalizing (e.g., substance use, antisocial disorder) or thought (e.g., schizophrenia, paranoid personality, bipolar) disorder that is uncontrolled or untreated
* Diagnosed with rheumatoid arthritis, osteoporosis, or cervical spine instability
* Hearing impairment (cognitive task uses auditory stimuli)
* Currently pregnant
* Current litigation related to a physical, health-related injury
* Whiplash injury in the past 3 months
* Oral injury, inflammation, or disease that causes the mouth or gums to bleed easily

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Recruitment | up to 6 months
  Average number of participants recruited/enrolled per month
Efficiency | 6 weeks
  Average battery duration
Latency | 6 weeks
  Average time between first lab assessment & first chiropractic session
Compliance | 6 weeks
  proportion of participants complying with pre-assessment lifestyle restrictions
Adherence | 6 weeks
  proportion of participants attending ≥80% of their chiropractic sessions
Tolerability | 6 weeks
  % of participants able to complete a given assessment
Retention | 6 weeks
  proportion of participants completing the trial
Acceptability | 6 weeks
  proportion of participant-rated & clinician-rated acceptability scores ≥3 in each domain
Data quality | 6 weeks
  % of acquisitions from a given assessment that are suitable for analysis

SECONDARY OUTCOMES:
Cognitive Flexibility | 6 weeks
  Modulation of executive function (i.e., cognitive flexibility) as indicated by changes in auditory switch task reaction time and decision error rate during gait
Gait | 6 weeks
  Modulation of gait as indicated by changes in the percentage of time spent in stance phase, load response, swing phase, single support, pre-swing, and initial swing.
Heart rate variability | 6 weeks
  Modulation of electrocardiography (ECG)-derived heart rate variability (HRV) during rest, stress, and recovery.
Pre-ejection period | 6 weeks
  Modulation of impedance cardiography (ICG)-derived pre-ejection period (PEP) during rest, stress, and recovery.
Secretory IgA | 6 weeks
  Modulation of immune activity as indicated by changes in salivary derived secretory immunoglobulin A (sIgA) levels at rest.
COMPASS-31 | 6 weeks
  Changes in self-reported autonomic function per the COMPASS-31 survey
PROMIS-29 | 6 weeks
  Changes in self-reported health related quality of life per the PROMIS-29 survey
PROMIS-Cog 8 | 6 weeks
  Changes in self-reported cognitive function per the PROMIS-Cognitive 8 survey
Perceived Stress Scale | 6 weeks
  Changes in self-reported stress per the Perceived Stress Scale (PSS).

CONTACTS AND LOCATIONS:
Overall Officials: Tyson Perez, DC, PhD, Principal Investigator — Life University
Locations (1):
- Dr. Sid E. Williams Center for Chiropractic Research, Marietta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT06208163/ICF_000.pdf